CLINICAL TRIAL: NCT02381639
Title: Impairment of Central Coherence in Restrictive Anorexia Nervosa: Single-center and Case-control Study
Brief Title: Impairment of Central Coherence in Restrictive Anorexia Nervosa (CoCA)
Acronym: CoCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC14_0301
Record Dates: First submitted 2015-02-10; First posted 2015-03-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2017-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Other): patients followed in the addiction service of the University Hospital of Nantes (consultations and / or hospitalizations) for restrictive anorexia nervosa
  Interventions: Behavioral: One interview of 90 minutes with a part of cognitive assessment and a part of self-assessment
- Healthy volunteers (Other): control subjects matched for age and sex with the patients
  Interventions: Behavioral: One interview of 90 minutes with a part of cognitive assessment and a part of self-assessment

INTERVENTIONS:
Behavioral: One interview of 90 minutes with a part of cognitive assessment and a part of self-assessment — The content of the assessment will be the same for all subjects and will consist of a part of cognitive assessment (National Reading Test, Rey Osterreich Complex Figure, Hayling Sentence Completion Task, verbal memory, digit sequencing, token motor task, verbal fluencies, symbol coding, tower of London) and self-assessment (Mini International Neuropsychiatric Interview, Beck Depression Inventory, State Trait Anxiety Inventory, Wender Utah Rating Scale, Adult Self-Report Scale Symptom Checklist, UPPS Impulsive Behavior Scale)

SUMMARY:
The current etiological pathological model of anorexia nervosa is poly-factorial involving individual genetic and psychological factors, in close interaction with environmental, family and socio-cultural factors.

Among these factors, this study focuses on the central coherence process (cognitive ability to integrate complex information into a comprehensive meaning), in the active phase of the disease. Therefore, patients followed in the addiction service of the Nantes University Hospital will perform neuropsychological tests assessing executive functions involved in the process of central coherence.

Impairment of central coherence process could act as a maintenance factor of the disease, particularly in connection with body dysmorphic disorder. The therapeutic perspectives acting on the central coherence process like cognitive remediation deserve to deepen knowledge on the cognitive profile of patients with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* For the patients :

  * Woman.
  * Aged of more than 15 years and 3 months.
  * Followed in the addiction service of the University Hospital of Nantes (consultations and / or hospitalizations) for Restrictive Anorexia Nervosa (according to the diagnostic criteria of DSM-IV-TR).
  * French language mastered.
  * Having signed the consent if major and if not the legal representatives have signed the consent (for minors).
* For the volunteers :

  * Women.
  * Aged of more than 15 years and 3 months.
  * French language mastered.
  * Having signed the consent if major and if not the legal representatives have signed the consent (for minors).

Exclusion Criteria:

* For the patients :

  * Man
  * Age under 15 years and 3 months old
  * Current Renutrition by nasogastric tube
  * Personal history of:

    * Head injury, neurodegenerative diseases, epilepsy unbalanced, unbalanced endocrine disorder, mental retardation
    * Support for current or past cognitive remediation
  * Opposition of the patient and / or his legal representatives if minor
  * Subject under legal guardianship
  * Current participation or in the past to pharmacological research protocol (time since the end of their participation in the protocol less than one year)
  * French language not mastered
* For the volunteers :

  * Man
  * Age under 15 years and 3 months old
  * Current Renutrition by nasogastric tube
  * Personal history of:

    * Eating disorders
    * Head injury, neurodegenerative diseases, epilepsy unbalanced, unbalanced endocrine disorder, mental retardation
    * Support for current or past cognitive remediation
  * Opposition of the volunteer and / or his legal representatives if minor
  * Subject under legal guardianship
  * Current participation or in the past to pharmacological research protocol (time since the end of their participation in the protocol less than one year)
  * French language not mastered

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Percentages for types I and III of the copy of the figure of Rey | 90 minutes

SECONDARY OUTCOMES:
Average scores for all cognitive and psychiatric tests | 90 minutes
Measure of relationships between average scores for all cognitive and psychiatric tests and socio-demographic and clinical data | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jennyfer CHOLET, Principal Investigator — Service d'Addictologie, CHU de Nantes, 44093 Nantes cedex 01, FRANCE
Locations (1):
- CHU de Nantes, Service d'Addictologie, Nantes, France